CLINICAL TRIAL: NCT04650204
Title: A Phase IV, Prospective, Open-Label, Parallel Study Evaluating the Effect of an Adjunctive Anti-Seizure Medication Using a Glutamatergic Modulator in Patients With Focal Epilepsy and High-Grade Glioma
Brief Title: Perampanel for the Reduction of Seizure Frequency in Patients With High-grade Glioma and Focal Epilepsy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The funding sponsor, EISAI, sold the US rights to the medication and can no longer provide it to patients for the study.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, William Tatum, DO, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 19-006286; NCI-2020-01290 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC2072 (Other: Mayo Clinic)
Record Dates: First submitted 2020-11-11; First posted 2020-12-02 (Actual); Results first posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-05

CONDITIONS: Intractable Epilepsy; Malignant Glioma; Seizure Disorder; WHO Grade 2 Glioma; WHO Grade 3 Glioma
MeSH Terms: conditions — Drug Resistant Epilepsy; Glioma; Epilepsy | interventions — Anticonvulsants; perampanel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (perampanel) (Experimental): Patients receive perampanel PO QD for 40 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Perampanel; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm B (ASD) (Active Comparator): Patients receive ASD per standard of care for 40 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Anticonvulsant Agent; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Anticonvulsant Agent — Given ASD
  Other Names: Anti-seizure agent; anticonvulsant; Anticonvulsant Agents; Anticonvulsants; antiepileptic; Antiepileptic Agent; Antiepileptics
  Arms: Arm B (ASD)
Drug: Perampanel — Given PO
  Other Names: E2007; Fycompa
  Arms: Arm A (perampanel)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase IV trial studies the side effects and how well perampanel works in reducing seizure frequency in patients with high-grade glioma and focal epilepsy. Perampanel is a drug used to treat seizures. Giving perampanel together with other anti-seizure drugs may work better in reducing seizure frequency in patients with high-grade glioma and focal epilepsy compared to alternate anti-seizure drugs alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Demonstrate the efficacy and safety of perampanel (PER) on seizure frequency in adult patients with biopsy-proven high-grade glioma and focal epilepsy compared with alternate anti-seizure drugs (ASDs).

SECONDARY OBJECTIVES:

I. To assess the change in neurocognitive function and brain magnetic resonance imaging (MRI) progression over the course of PER treatment with a daily dose of 4 mg (up to -8mg) in patients with biopsy-proven high-grade glioma and focal epilepsy compared with alternate ASDs.

II. To identify a biomarker-specific response to seizure-reduction in patients treated with PER in patients with a biopsy-proven high-grade glioma (i.e., IDH-mutant versus [vs] wildtype).

OUTLINE: Patients are assigned to 1 of 2 groups.

GROUP A: Patients receive perampanel orally (PO) once daily (QD) for 40 weeks in the absence of disease progression or unacceptable toxicity.

GROUP B: Patients receive ASD per standard of care for 40 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* The subject, or the subject's legally acceptable representative is willing to participate in a clinical trial, provides written informed consent, and subject provides written assent, as required by the Mayo Clinic Institutional Review Board (IRB) policy involving human subjects. In the event of subject lacking the capacity or losing the ability to consent, consent will be deferred to subject's legally acceptable representative
* Subjects that meet the following diagnostic criteria:

  * Patients with established clinical diagnoses of biopsy-proven high-grade glioma (grade II or above) and epilepsy refractory to at least 1, drug with a seizure frequency of at least 1 seizure episode per month prior to baseline visit
* Subjects with body weight of >= 40 kg and =< 125 kg at screening
* Adults age 18 and older

Exclusion Criteria:

* Subject has serious cardiac, respiratory, renal, gastrointestinal, hematologic, or other medical condition as determined by the investigator to potentially interfere with the study
* Subjects with glioblastoma not following Stupp protocol for treatment of glioblastoma
* History of status epilepticus in the 6 months prior to screening or a history of seizure clusters progressing to status epilepticus
* Past medical history of drug and/or alcohol abuse
* Pregnant or breast-feeding
* Subjects treated with PER prior to baseline
* Prior felony conviction disclosed by the patient or previously stated in medical record
* History of violent behavior
* Clinically significant laboratory abnormality at screening or baseline visits, as determined by the investigators
* Use of an investigational drug or device within 20 days prior to treatment day 1
* Repeated radiation therapy for tumor regrowth
* Subjects that plan to undergo tumor resection on or after baseline visit
* Uncontrolled psychiatric disorder at baseline
* Subjects who report active suicidal attempts or suicidality including subjects with a history of suicide attempts or suicidality determined to be clinically significant by investigators at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-12-04 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Tatum, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A (Perampanel) | Arm B (ASD)
Started | 3 | 1
Completed | 1 | 0
Not Completed | 2 | 1
Not completed — Study was Terminated | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Perampanel) | Arm B (ASD) | Total
Number analyzed (Participants) | 3 | 1 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 4
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 1 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With a High-grade Glioma Who Achieve a > 50% Reduction in Focal Seizures With Perampanel (PER) 4 mg Daily After Failing 1 or More Anti-seizure Drugs (ASDs)
Description: Will compare seizure frequency before and 3 months after treatment with monotherapy and adjunctive PER and use descriptive statistics to demonstrate differences in responders. A P-value < 0.05 will be used to reflect statistical significance.
Time Frame: At 3 months
Population: 1 participant was randomized to Arm B, but did not complete the 3 month follow-up due to study termination. In Arm A, only 2 participants met the study 3 month mark prior to study termination.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Perampanel) | Arm B (ASD)
Number analyzed (Participants) | 2 | 0
Participants | 1 |

2. Primary Outcome: Number of Patients With a High-grade Glioma Who Achieve a > 50% Reduction in Focal Seizures With PER 4 mg Daily After Failing 1 or More ASDs
Description: Will compare seizure frequency before and 6 months after treatment with monotherapy and adjunctive PER and use descriptive statistics to demonstrate differences in responders. A P-value < 0.05 will be used to reflect statistical significance.
Time Frame: At 6 months
Population: 1 participant was randomized to Arm B, but did not complete the 6 month follow-up due to study termination. In Arm A, only 1 participant met the study 6 month mark prior to study termination.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Perampanel) | Arm B (ASD)
Number analyzed (Participants) | 1 | 0
Participants | 1 |

3. Primary Outcome: Number of Participants Alive at 3 Months With High-grade Glioma Treated With PER
Description: Chi-square and Student T-test will be used to measure differences in assessment and change during the study period.
Time Frame: At 3 months
Population: 1 participant was randomized to Arm B, but did not receive PER treatment. In Arm A, only 2 participants met the study 3 month mark prior to study termination.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Perampanel) | Arm B (ASD)
Number analyzed (Participants) | 2 | 0
Participants | 2 |

4. Primary Outcome: Decline in Neuropsychological Function
Description: Chi-square and Student T-test will be used to measure differences in assessment and change during the study period.
Time Frame: At 6 months
Population: The study was terminated due to the funding sponsor no longer being able to provide study medication. Data for this outcome measure was not collected nor analyzed.
Arm/Group | Arm A (Perampanel) | Arm B (ASD)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from a baseline to end of study participation for approximately 12 months on all participants.
Arm/Group | Arm A (Perampanel) | Arm B (ASD)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/1
Other Adverse Events (participants affected / at risk) | 2/3 | 0/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Perampanel) (N=3) | Arm B (ASD) (N=1)
Imbalance & problems with coordination (Nervous system disorders) | 1 (1) | 0 (0)
Urinary Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Valproic acid Toxicity (General disorders) | 1 (1) | 0 (0)
Headaches (Nervous system disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Study was terminated due to the funding sponsor(EISAI) sold the US rights to the medication and can no longer provide it to patients for the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-23): https://cdn.clinicaltrials.gov/large-docs/04/NCT04650204/Prot_SAP_000.pdf